CLINICAL TRIAL: NCT06439082
Title: A Phase III, Multicenter, Randomized, Placebo Controlled, Double-blind Study to Assess Efficacy and Safety of Crizanlizumab (5 mg/kg) Versus Placebo, With or Without Hydroxyurea/Hydroxycarbamide Therapy, in Adolescent and Adult Sickle Cell Disease Patients With Frequent Vaso-Occlusive Crises
Brief Title: A Study to Investigate the Efficacy and Safety of Crizanlizumab (5 mg/kg) Compared With Placebo in Adolescent and Adult Sickle Cell Disease Patients Who Experience Frequent Vaso-Occlusive Crises (SPARKLE)
Acronym: SPARKLE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSEG101A2303
Expanded Access: NCT03720626 (Available)
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; SCD; SEG101; Crizanlizumab; Hydroxyurea/ Hydroxycarbamide Therapy; Vaso-Occlusive Crises; Sickle Cell Anemia; blood disorders; hemoglobin; red blood cells; sickle-like shape; mutation in hemoglobin gene; sickle-cell trait; sickle-cell crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hematologic Diseases; Sickle Cell Trait | interventions — crizanlizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crizanlizumab (SEG101) at 5.0 mg/kg (Experimental): Participants receive Crizanlizumab (SEG101) at 5.0 mg/kg and standard of care.
  Interventions: Biological: Crizanlizumab
- Placebo (Placebo Comparator): Participants receive the placebo drug and standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Crizanlizumab — Crizanlizumab is supplied in single use 10 mL glass vials at a concentration of 10 mg/mL. One vial contains 100 mg of crizanlizumab. This is a concentrate for solution for IV infusion.
  Other Names: SEG101, Adakveo®, Ryverna®
  Arms: Crizanlizumab (SEG101) at 5.0 mg/kg
Drug: Placebo — Placebo is supplied in single use 10 mL glass vials at a concentration of 0 mg/mL. This is a concentrate for solution for IV infusion.
  Arms: Placebo

SUMMARY:
A phase III, multi-center, randomized, placebo-controlled, double-blind study to assess efficacy and safety of crizanlizumab (5 mg/kg) versus placebo, with or without hydroxyurea/hydroxycarbamide therapy, in adolescent and adult Sickle Cell Disease patients with frequent vaso-occlusive crises.

DETAILED DESCRIPTION:
Study CSEG101A2303 (SPARKLE) is a Phase III, multicenter, randomized, double-blind study to assess efficacy and safety of crizanlizumab 5 mg/kg versus placebo, with or without hydroxyurea/ hydroxycarbamide therapy (HU/HC), in Sickle Cell Disease patients aged 12 years and older with frequent vaso-occlusive crises (4-12 events in 12 months prior to the screening visit).

Participants will be randomized in a 2:1 ratio to the crizanlizumab 5 mg/kg or placebo treatment arm. Central randomization will be stratified by concomitant HU/HC usage (yes/no) and region (South America, North America, and sub-Saharan Africa) at baseline.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must be aged 12 years and older on the day of signing informed consent. Adolescents include participants aged 12 to <18 years old and adults include participants aged 18 years and older.
2. Confirmed diagnosis of SCD by Hb electrophoresis or high-performance liquid chromatography (HPLC) (performed locally or by central laboratory if not available locally). All SCD genotypes are eligible.
3. Experienced 4 to 12 VOCs (refer to Section 8.3.1 for study definition of VOC) that are HCP-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) within the 12 months prior to the screening visit. Baseline VOCs are determined by medical history and are required to be documented at source.
4. If the participant is on HU/HC, they must be taking it for at least 6 months and at stable dose for at least 3 months prior to the Screening visit and plan to continue taking it at the same dose and schedule until at least the participant has reached 52 weeks of the planned study treatment. Participants who have initiated HU/HC 6-12 months prior to the screening visit must have evidence of insufficient control of acute pain despite initiation. These participants must have a cumulative of 4-12 VOCs in the 12 months prior to the screening period, with at least 2 during the last 6 months while on HU/HC. If receiving erythropoietin stimulating agent, the participant must have been receiving the drug for at least 6 months prior to screening visit and plan to continue taking the drug at the same dose and schedule until the participant has reached 52 weeks of the planned study treatment.

Participants who have not been receiving HU/HC, and/or erythropoietin stimulating agent must not have received it for at least 6 months prior to screening visit.

Key Exclusion Criteria:

1. Fewer than 4 or more than 12 VOCs that are HCP-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) within the 12 months prior to screening visit as determined by medical history and documented at source.
2. History of stem cell transplant and/or gene therapy.
3. Received blood products within 30 days prior to Week 1 Day 1 dosing.
4. Any documented history of a clinical stroke or intracranial hemorrhage, or an uninvestigated neurologic finding within the past 12 months before screening visit. Silent infarct only present on imaging is not excluded.
5. Participating in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes) and/or planning to undergo an exchange transfusion during the duration of the study; episodic transfusion in response to worsened anemia or VOC is permitted.
6. Contraindication or hypersensitivity to any drug or metabolites from similar class as study drug or to any excipients of the study drug formulation. History of severe hypersensitivity reaction to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2029-03-23 (Estimated); Study Completion 2030-04-19 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of VOCs that are healthcare professional (HCP)-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) in each treatment arm | 1 year
  Vaso oclusive crisis (VOC) is defined as a pain crisis (acute onset of pain for which there is no other medically determined explanation other than vaso-occlusion) lasting for at least 4 hours which is treated as per local guidelines with standard of care therapy used to treat VOC. Acute chest syndrome (ACS), priapism and hepatic or splenic sequestration will be considered VOC in this study.
  VOCs included are those HCP-managed in a healthcare facility and HCP-managed via remote consultation.
  Annualized rate of VOC events = (Number of VOC events * 365)/(number of days in the observation period).
  Observation period = time from date of randomization to minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-Glutamine (or other therapies such as Voxelotor and erythropoietin therapies to treat SCD and/or to prevent/reduce VOCs), date of randomization + 365 days).

SECONDARY OUTCOMES:
The annualized rate of all VOCs including VOCs that are HCP-managed (either at a health care facility or via remote consultation) as well as those that are self-managed without recommendations from HCP during the event in each treatment arm | 1 year
  VOCs can be categorized as those HCP-managed in a healthcare facility, HCP-managed via remote consultation, or self-managed without recommendations from HCP during the event.
  Annualized rate of VOC events = (Number of VOC events * 365)/(number of days in the observation period).
  To capture VOC events that are self-managed, and in order to avoid VOC recall bias and to make sure the pain events are captured in real-time, a cloud-based application will be used and setup an account for each participant.
Annualized rate of VOC by subtype of management in each treatment arm over the planned 52-week period. | 1 year
  Vaso oclusive crisis (VOC) is defined as a pain crisis lasting for at least 4 hours which is treated as per local guidelines with standard of care therapy. Acute chest syndrome (ACS), priapism and hepatic or splenic sequestration will be considered VOC in this study.
  VOCs can be categorized as those HCP-managed in a healthcare facility, HCP-managed via remote consultation, or self-managed without recommendations from HCP during the event.
  Annualized rate of VOC is the number of VOC events during a year period.
The time to first VOC that is HCP-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) between treatment arms. | 1 year
  VOC is defined as a pain crisis lasting for at least 4 hours which is treated as per local guidelines with standard of care therapy. ACS, priapism and hepatic or splenic sequestration will be considered VOC in this study.
  VOCs included are those HCP-managed in a healthcare facility and HCP-managed via remote consultation.
  Time to first occurrence of VOC that is HCP-managed (either at a health care facility or via remote consultation) is defined as the time from the date of randomization to the date of the first occurrence of the VOC.
Proportion of participants free from VOCs that are HCP-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) in each treatment arm over the planned 52-week treatment period. | 1 year
  To assess the number of participants free from VOCs leading to healthcare visit.
  VOC is defined as a pain crisis lasting for at least 4 hours which is treated as per local guidelines with standard of care therapy. ACS, priapism and hepatic or splenic sequestration will be considered VOC in this study. A participant is free from VOC if they do not have a VOC crisis.
Duration of VOCs that are HCP-managed (including VOCs leading to management at a health care facility or those managed via remote consultation) in each treatment arm over the planned 52-week treatment period. | 1 year
  VOC is defined as a pain crisis lasting for at least 4 hours which is treated as per local guidelines with standard of care therapy. ACS, priapism and hepatic or splenic sequestration will be considered VOC in this study.
  Duration of HCP-managed VOC is defined as end date of the VOC - start date of the VOC + 1 day.
Number of participants with anti-SEG101 (crizanlizumab) antibodies (any time) | 2 years
  Immunogenicity: measurement of anti-drug antibodies (ADA) to crizanlizumab.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 2 years
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs), and laboratory results qualifying and reported as AEs.
Absolute change from baseline in hemoglobin | Baseline, 2 years
  Assessment of safety of SEG101

CONTACTS AND LOCATIONS:
Locations (17):
- United States (13):
  - University Of Alabama, Birmingham, Alabama
  - Childrens National Hospital, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - Augusta University Georgia, Augusta, Georgia
  - WCG Sonar Clinical Research, Riverdale, Georgia
  - Norton Children s Hospital, Louisville, Kentucky
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Southern Specialty Research, Flowood, Mississippi
  - Childrens Hospital at Montefiore, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Spoknwrdclinicaltrials, Easton, Pennsylvania
  - U of TX Health Science Ct, Houston, Texas
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Montería
- Novartis Investigative Site, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com